CLINICAL TRIAL: NCT04564300
Title: Influence of Oral Contraceptive Use on Recovery in Trained Women
Brief Title: The Influence of Oral Contraceptive Use on Muscle Recovery
Acronym: OC-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OC-R
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Recovery; Oral Contraceptive Use

STUDY DESIGN:
Intervention Model Description: We will compare the recovery in a group of oral contraceptive users to a group of women not using oral contraceptives
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral contraceptive users (Experimental)
  Interventions: Procedure: Training
- Non-oral contraceptive users (Active Comparator)
  Interventions: Procedure: Training

INTERVENTIONS:
Procedure: Training — Both groups will perform a standardized training protocol

SUMMARY:
There is still no one who has studied how oral contraceptive use affects recovery in trained women after repeated high-intensity workouts. Consequently, a well-controlled study is needed.

The project is designed as a controlled cohort study, where 20 oral contraceptive users will be compared with 20 non-users. After initial preliminary examination and habituation to the test procedures, the subjects will start the intervention in week 2 of their menstrual cycle / active contraceptive pill cycle. Before and 3h, 24h and 48h after 3 intense strength training sessions performed 2 days in a row, blood samples will be taken, muscle soreness measured and performance tests performed. The day before the first training session and over the 4 trial days, the subjects will receive a standardized diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-30
* Regular training minimum. 4 times a week (1≤ times strength training, 1≤ times endurance training / interval training or interval-based sports. If the interest in participation is greater than necessary, we will prioritize people who perform strength training at least twice a week)

Exclusion Criteria:

* Irregular menstruation over the last 6 months (shorter than 24 days or longer than 35 days cycle)
* Used birth control pills for less than 6 months
* Non-birth control pill users must not have used birth control pills, IUDs, birth control pills, or mini- pills for a maximum of 1 month during the last 6 months and not within the last 3 months up to the trial. .
* Injuries / pain in the lower body, which prevents participation in intense strength training
* Medication consumption that may affect protein metabolism and inflammatory parameters.
* Diabetes
* Smoking
* Unstable weight / major weight loss (weight fluctuations of more than 5 kg in the last six months)
* Eating disorder
* Pregnancy
* Cannot read or understand Danish

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Changes in maximal knee extensor strength and Rate of force development | Before, 3 hours , 24 hours and 48 hours after training
  Measured in a Humac Norm dynamometer

SECONDARY OUTCOMES:
Changes in Jumping performance | Before, 3 hours , 24 hours and 48 hours after training.
  Jump height
Changes in Jumping performance | Before, 3 hours , 24 hours and 48 hours after training.
  Power
Changes in Jumping performance | Before, 3 hours , 24 hours and 48 hours after training.
  modified reactive strength index
Changes in Jumping performance | Before, 3 hours , 24 hours and 48 hours after training.
  leg stiffness
Changes in Wingate performance | Before, 3 hours , 24 hours and 48 hours after training.
  Peak power and average power
Changes in Yoyo-intermittent recovery 1 performance | Before, and 48 hours after training.
  total length covered in the yo-yo test
Changes in Leg press performance | Before, 3 hours , 24 hours and 48 hours after training.
  Total reps performed at 80% of 1RM
Changes training volume | Before, 3 hours , 24 hours and 48 hours after training.
  total volume performed during training (i.e set x reps x working weight)
Differences in knee laxity | Baseline
  Measured with a Lachmeter
Changes in muscle soreness (VAS-score) | Before, 3 hours , 24 hours and 48 hours after training
  Subjects will raise and sit on a chair and immediately after answer a VAS-score (100mm line, from worst pain ever, to no pain at all.)
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  estradiol
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  testosterone
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  sex hormone-binding globulin
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  progesterone
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  follicle-stimulating hormone
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  luteinizing hormone
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  Creatine kinase
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  Lactate dehydrogenase
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  Myoglobin
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  Cortisol
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  C-reactive protein
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  tumor necrosis factor
Blood analysis: Sex hormones, cortisol, inflammatory markers and markers of muscle damage | Before, 3 hours , 24 hours and 48 hours after training
  IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No